CLINICAL TRIAL: NCT00000736
Title: Safety and Efficacy of Zidovudine for Asymptomatic HIV-Infected Individuals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 019; 10995 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine if treatment with zidovudine (AZT) will delay or prevent the onset of AIDS or AIDS related complex (ARC) in individuals infected with HIV but who do not have symptoms of AIDS or ARC. Also, to compare the dose of AZT found to be useful in AIDS and severe ARC with a lower dose to see if side effects can be reduced.

Results from several studies show that a high percentage of people infected with HIV will eventually develop AIDS or ARC unless an effective treatment is found. Because AZT is known to prolong survival in patients with AIDS or severe ARC and has acceptable toxicity in advanced disease, it is reasonable to try it in less advanced cases.

DETAILED DESCRIPTION:
Results from several studies show that a high percentage of people infected with HIV will eventually develop AIDS or ARC unless an effective treatment is found. Because AZT is known to prolong survival in patients with AIDS or severe ARC and has acceptable toxicity in advanced disease, it is reasonable to try it in less advanced cases.

Patients entered in the study are randomly assigned to one of two doses of AZT or to placebo (inactive medication). Patients take 3 capsules 5 times a day (every 4 hours from 8 am until 12 pm).

The capsules contain either AZT or placebo and are identical in appearance so that neither patient nor physician knows which treatment the patient is receiving. The higher dose corresponds to the dose found to be useful in patients with AIDS or severe ARC. Patients visit the clinic every 2 weeks for the first 16 weeks, then once a month after that for evaluation. Treatment will continue until the results from the study have been analyzed, which could be as long as 3 years. If side effects occur, the dose of study medication will be decreased or temporarily stopped. If the side effects are severe, then study medication will be stopped permanently.

AMENDED: Effective with Version 4 (900226), dosing for ALL patients on Phase 2 study drug, regardless of CD4+ substudy, will proceed as open-label AZT. Original treatment assignments employed in the > 500 cells/mm3 substudy during the period from August 16, 1989 through the release of this new version. Also, toxicity management and dose modification of AZT for patients receiving Phase 2 study drug have been changed.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* Be HIV seropositive and asymptomatic.
* Have normal neurologic exam as defined by the Micro Neuro-AIDS assessment.

Concurrent Medication

* Required: Prophylaxis for Pneumocystis carinii pneumonia (PCP). Aerosolized pentamidine is preferred but if not possible, Trimethoprim / sulfamethoxazole 1 DS tablet per day or Dapsone 50 - 100 mg per day is allowed.

Exclusion Criteria

* Active drug or alcohol abuse sufficient to prevent adequate compliance with study therapy in the investigator's opinion.

Co-existing Condition:

Patients with the following diseases or conditions are excluded:

* Hemophilia.
* Oral candida infection documented by morphology or by response to antifungal therapy within 2 years of study entry.
* Oral hairy leukoplakia at any time prior to study entry.
* Herpes zoster infection (including single dermatome infection) within 2 years of study entry.
* Active diarrhea as defined by 3 or more liquid stools per day.
* Temperature > 37.8 degrees C.
* Grade 1 impairment on two or more items (mild AIDS dementia complex) in the ACTG Micro Neuro-AIDS Assessment.
* Prior history of malignancy other than cutaneous basal cell carcinomas or cervical carcinoma in situ.

Patients with the following are excluded from entry:

* AIDS or AIDS-related complex defining symptoms.
* Significant, chronic underlying medical illnesses which would impair continuous participation in this 3-year clinical trial.
* Hemophilia.

Prior Medication: Excluded:

* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP).
* Other experimental medications.
* Excluded within 60 days of study entry:
* Antiretroviral drugs or immunomodulators (biologic response modifiers).
* Excluded within 120 days of study entry:
* Systemic corticosteroids.

Prior Treatment: Excluded within 3 months of study entry:

* Blood transfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volberding P, Study Chair
Locations (43):
- United States (43):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Children's Hosp of San Francisco, San Francisco, California
  - San Francisco AIDS Clinic, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Volberding PA, Lagakos SW, Grimes JM, Stein DS, Balfour HH Jr, Reichman RC, Bartlett JA, Hirsch MS, Phair JP, Mitsuyasu RT, et al. The duration of zidovudine benefit in persons with asymptomatic HIV infection. Prolonged evaluation of protocol 019 of the AIDS Clinical Trials Group. JAMA. 1994 Aug 10;272(6):437-42. PMID 7913730
- [Background] Choi S, Lagakos SW, Schooley RT, Volberding PA. CD4+ lymphocytes are an incomplete surrogate marker for clinical progression in persons with asymptomatic HIV infection taking zidovudine. Ann Intern Med. 1993 May 1;118(9):674-80. doi: 10.7326/0003-4819-118-9-199305010-00003. PMID 8096373
- [Background] Volberding PA, Lagakos SW, Grimes JM, Stein DS, Rooney J, Meng TC, Fischl MA, Collier AC, Phair JP, Hirsch MS, et al. A comparison of immediate with deferred zidovudine therapy for asymptomatic HIV-infected adults with CD4 cell counts of 500 or more per cubic millimeter. AIDS Clinical Trials Group. N Engl J Med. 1995 Aug 17;333(7):401-7. doi: 10.1056/NEJM199508173330701. PMID 7616988
- [Background] Vella S, Giuliano M, Dally LG, Agresti MG, Tomino C, Floridia M, Chiesi A, Fragola V, Moroni M, Piazza M, et al. Long-term follow-up of zidovudine therapy in asymptomatic HIV infection: results of a multicenter cohort study. The Italian Zidovudine Evaluation Group. J Acquir Immune Defic Syndr (1988). 1994 Jan;7(1):31-8. PMID 7903380
- [Background] Volberding PA, Lagakos SW, Koch MA, Pettinelli C, Myers MW, Booth DK, Balfour HH Jr, Reichman RC, Bartlett JA, Hirsch MS, et al. Zidovudine in asymptomatic human immunodeficiency virus infection. A controlled trial in persons with fewer than 500 CD4-positive cells per cubic millimeter. The AIDS Clinical Trials Group of the National Institute of Allergy and Infectious Diseases. N Engl J Med. 1990 Apr 5;322(14):941-9. doi: 10.1056/NEJM199004053221401. PMID 1969115
- [Background] Volberding P. The value of the CD4+ count of 500 cells/microliters. Drugs. 1995;49 Suppl 1:4-8; discussion 38-40. doi: 10.2165/00003495-199500491-00004. PMID 7614901
- [Background] Lenderking WR, Gelber RD, Cotton DJ, Cole BF, Goldhirsch A, Volberding PA, Testa MA. Evaluation of the quality of life associated with zidovudine treatment in asymptomatic human immunodeficiency virus infection. The AIDS Clinical Trials Group. N Engl J Med. 1994 Mar 17;330(11):738-43. doi: 10.1056/NEJM199403173301102. PMID 7906386
- [Background] Wu AW, Rubin HR, Mathews WC, Ware JE Jr, Brysk LT, Hardy WD, Bozzette SA, Spector SA, Richman DD. A health status questionnaire using 30 items from the Medical Outcomes Study. Preliminary validation in persons with early HIV infection. Med Care. 1991 Aug;29(8):786-98. doi: 10.1097/00005650-199108000-00011. PMID 1875745
- [Background] Jacobson MA, Gundacker H, Hughes M, Fischl M, Volberding P. Zidovudine side effects as reported by black, Hispanic, and white/non-Hispanic patients with early HIV disease: combined analysis of two multicenter placebo-controlled trials. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Jan 1;11(1):45-52. doi: 10.1097/00042560-199601010-00006. PMID 8528732